CLINICAL TRIAL: NCT00828178
Title: A Randomized, Double-blind, Placebo-controlled, Clinical Trial of Omega-3-polyunsaturated Fatty Acids in Subjects With SLE.
Brief Title: Efficacy of Fish Oil in Lupus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michelle Petri M.D.,MPH (Other)
Responsible Party: Sponsor-Investigator, Michelle Petri M.D.,MPH, Principal investigator, Johns Hopkins University
Organization: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00023813
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; atherosclerosis; omega-3
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Atherosclerosis | interventions — Docosahexaenoic Acids; Omacor; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 (Active Comparator): 3 g of Omega-3 (1.8 g eicosapentaenoic acid, 1.2 g docosahexaenoic acid ethyl esters); flow-mediated dilation of the brachial artery
  Interventions: Drug: Omega-3; Device: flow-mediated dilation of the brachial artery
- corn starch (Placebo Comparator): corn starch; flow-mediated dilation of the brachial artery
  Interventions: Device: flow-mediated dilation of the brachial artery; Other: corn starch

INTERVENTIONS:
Drug: Omega-3 — Omega-3-acid ethyl esters (Lovaza) 3 gram once a day for 12 weeks
  Other Names: Lovaza
  Arms: Omega-3
Device: flow-mediated dilation of the brachial artery — flow-mediated dilation of the brachial artery measurement at baseline and after 12 weeks
Other: corn starch — 3 capsules qd for 12weeks
  Arms: corn starch

SUMMARY:
The investigators hypothesize that low-dose dietary supplementation with omega-3 fish oil will improve disease activity and endothelial function in Systemic Lupus Erythematosus (SLE) patients.

DETAILED DESCRIPTION:
Patients with SLE have a fifty-fold increased risk of myocardial infarction. This risk is not totally explained by traditional cardiovascular risk factors. In a previous double-blind study of atorvastatin in SLE, there was no reduction in surrogate measures of coronary artery disease (coronary calcium, coronary IMT, carotid plaque) and no effect on inflammatory markers such as ICAM, VCAM, IL-6 and CRP. We need to find novel approaches to reduce coronary artery disease in SLE. In a preliminary study, omega-3 was shown to improve flow mediated dilation of the brachial artery, oxidative stress and disease activity in lupus patients. In this study we will determine if omega-3 improves brachial artery flow dilation, disease activity and other vascular inflammatory markers (IL-6, s-VCAM-1, s-ICAM-1) in SLE, in a double-blind placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of SLE are eligible.
* Patients must be 18 years of age or older and able to give informed consent.

Exclusion Criteria:

* SLE patients who are allergic to fish oil or any omega 3 product.
* Patients who are pregnant or are planning to become pregnant or are nursing.
* Omega-3 use within the previous 6 weeks of enrollment.
* Use of warfarin or heparin.
* Patients who have coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Petri, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Lupus Center, Johns Hopkins University, Baltimore, Maryland
  - The Johns Hopkins Lupus Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manzi S, Meilahn EN, Rairie JE, Conte CG, Medsger TA Jr, Jansen-McWilliams L, D'Agostino RB, Kuller LH. Age-specific incidence rates of myocardial infarction and angina in women with systemic lupus erythematosus: comparison with the Framingham Study. Am J Epidemiol. 1997 Mar 1;145(5):408-15. doi: 10.1093/oxfordjournals.aje.a009122. PMID 9048514
- [Result] Duffy EM, Meenagh GK, McMillan SA, Strain JJ, Hannigan BM, Bell AL. The clinical effect of dietary supplementation with omega-3 fish oils and/or copper in systemic lupus erythematosus. J Rheumatol. 2004 Aug;31(8):1551-6. PMID 15290734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 106 patients were consented and 87 were randomized. Patients were part of the Hopkins Lupus Cohort seen quarterly.
Pre-assignment Details: Some of patients were excluded before being randomized for several reasons including "change of mind by patient, became pregnant, diagnosed with breast ca". Therefore a total of 87 patients started the trial.
Groups:
- Fish Oil: fish oil 3 g of Omega-3 (1.8 g eicosapentaenoic acid, 1.2 g docosahexaenoic acid ethyl esters) daily
- Placebo: Placebo (corn starch) once daily
Period: Overall Study
Arm/Group | Fish Oil | Placebo
Started | 42 | 45 (Eighty seven participants were randomized.)
Completed | 42 | 43 (Two patients did not complete the study.)
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Fish Oil: 3 g of Omega-3 (1.8 g eicosapentaenoic acid, 1.2 g docosahexaenoic acid ethyl esters)
- Placebo: corn starch
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Placebo | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 45 | 87
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (10.6) | 45.5 (10.8) | 47.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 42 | 45 | 87

OUTCOME MEASURES:

1. Primary Outcome: Effect on Brachial Artery Flow Dilation by Omega-3 Versus Placebo.
Description: The assessment measured mean brachial artery diameter at pre-treatment(baseline) and post-treatment (after 12 weeks).
Time Frame: 12 weeks
Population: Patients who successfully completed the trial.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Omega-3: 3 g of Omega-3 (1.8 g eicosapentaenoic acid, 1.2 g docosahexaenoic acid ethyl esters)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 42 | 43
cm
  Post-treatment baseline diameter | 0.32 (0.04) | 0.33 (0.06)
  Pre-treatment baseline diameter | 0.32 (0.06) | 0.33 (0.06)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Statistical analysis system (SAS) software was used (SAS Institute Inc. Cary, North Carolina, SAS 9.2). Baseline demographic and clinical characteristics were summarized using appropriate descriptive statistics and compared across treatment groups using Chi-square. Two-sample t tests were used in the statistical analysis of the FMD outcomes. ANCOVA was used to compare the groups with respect to changes in clinical variables adjusting for baseline values; Test type: Superiority or Other; p = 0.87, t-test, 2 sided

2. Secondary Outcome: Effect of Omega-3 Versus Placebo on Disease Activity in SLE.
Description: The assessment measured change in disease activities using SELENA-SLEDAI (Systemic Lupus Erythematosus Disease Activity Index Selena Modification - range 0-105) and PGA (Physician Global Assessment - range 0-3) comparing pre-treatment(baseline) vs post-treatment (after 12 weeks).
  SELENA-SLEDAI - range 0-105, high score indicates high disease activity - weighted sum of sub-scale is used as total score.
  PGA - range 0-3, high score indicates high disease activity.
Time Frame: pre-treatment(baseline) and post-treatment (after 12 weeks)
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Placebo (cornstarch)
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 42 | 43
Units on a scale
  SELENA-SLEDAI | 1.5 (2) | 1.5 (2.5)
  PGA | 0.49 (0.52) | 0.41 (0.49)
Statistical Analysis 1: Comparison: Omega-3 vs Placebo; Test type: Superiority or Other; p = 0.1801, t-test, 2 sided — This Statistical Analysis applies category SELENA-SLEDAI

3. Secondary Outcome: Effect on Markers of Inflammation: ICAM and VCAM by Omega-3 Versus Placebo.
Description: The inflammatory markers (sICAM-1 and sVCAM-1) were assessed and compared before and after treatment. change from baseline were reported.
Time Frame: pre-treatment(baseline) and post-treatment (after 12 weeks)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Omega-3 | Placebo
Number analyzed (Participants) | 42 | 43
ng/ml
  sICAM-1 | -1.61 (40.27) | -5.56 (48.74)
  sVCAM-1 | -17.52 (101.65) | 26.57 (135.98)

ADVERSE EVENTS:
Arm/Group | Omega-3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No